CLINICAL TRIAL: NCT04865133
Title: Efficacy and Safety of COVID-19 Vaccine in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 21-001818; NCI-2021-03137 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-04-22; First posted 2021-04-29 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: COVID-19 Infection; Malignant Solid Neoplasm
MeSH Terms: conditions — COVID-19 | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection, medical record): Patients undergo blood sample collection at baseline (prior to first COVID-19 vaccination), prior to second vaccination, 1, 6, and 12 months after the last vaccination. Patients receiving a booster vaccine will undergo blood collection prior to and 1-3 months after vaccination. Patients who receive the types of COVID-19 vaccines that do not require the second injection skip blood sample collection at this time point. This study will collect information regarding the type of COVID-19 vaccine received, date of vaccine injection, and any side effects associated with the COVID-19 vaccine that trial participant encountered. This study will also review the medical record for outcomes and information related to the blood testing.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Medical record reviewed

SUMMARY:
This study gathers information about how a cancer patient responds to COVID-19 vaccine during cancer treatment compared to healthy individuals. The information gained may help determine how effective currently available COVID-19 vaccines are in cancer patients receiving chemotherapy and learn more regarding how long an immune response will last compared to healthy individuals.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the antibody response to COVID-19 vaccine after vaccination. II. To assess the adverse events of COVID-19 vaccines in cancer patients. III. To determine the incidence and severity of COVID-19 infection after the vaccination.

OUTLINE:

Patients undergo blood sample collection at baseline (prior to first COVID-19 vaccination), prior to second vaccination, 1, 6, and 12 months after the last vaccination. Patients receiving a booster vaccine will undergo blood collection prior to and 1-3 months after vaccination. Patients who receive the types of COVID-19 vaccines that do not require the second injection skip blood sample collection at this time point. This study will collect information regarding the type of COVID-19 vaccine received, date of vaccine injection, and any side effects associated with the COVID-19 vaccine that trial participant encountered. This study will also review the medical record for outcomes and information related to the blood testing.

ELIGIBILITY:
Inclusion Criteria:

* Willing to receive COVID-19 vaccination as per standard of care or has already received one or both COVID-19 vaccine injections as long as it has not been longer than three months since their second injection (or the only injection if they receive the types of COVID019 vaccines that do not require the second injection)
* Willing and able to provide research blood samples
* Capable of providing valid informed consent
* For cancer patient cohort:

  * Male or female age >= 18 years
  * Histologically confirmed solid malignancy on or will be starting on systemic cytotoxic chemotherapy
* For healthy individual cohort:

  * Male or female age >= 18 years
  * No history of active malignancy =< 3 years
* EXCEPTIONS: Adequately treated non-melanotic skin cancer (adequate wound healing is required prior to study entry) or carcinoma-in-situ of the cervix
* NOTE: If there is a history of prior solid tumor malignancy, it must have been treated curatively with no evidence of recurrence =< 3 years
* PATIENTS WITH PREVIOUS COVID-19 INFECTION: Willing and able to provide research blood samples
* PATIENTS WITH PREVIOUS COVID-19 INFECTION: Capable of providing valid informed consent
* PATIENTS WITH PREVIOUS COVID-19 INFECTION: Male or female age >= 18 years
* PATIENTS WITH PREVIOUS COVID-19 INFECTION: Previous history of COVID-19 infection with positive SARS-CoV-2 ribonucleic acid (RNA) by polymerase chain reaction (PCR) or anti-SARS-CoV-2 nucleocapsid antibody

Exclusion Criteria:

* Immunocompromised patients including patients known to be human immunodeficiency virus (HIV) positive or those on immunosuppressive therapy other than chemotherapy in the judgment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with cancer on or will be starting on systemic cytotoxic chemotherapy for their cancer and healthy individuals who will receive COVID-19 vaccine
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Antibody response to COVID-19 vaccine after vaccination in cancer patients and health individuals | Up to 12 months
  Wilcoxon rank sum test will be used to compare between baseline and other 3 time points (before the second vaccination, 3 months, and 12 months after the second vaccination).

SECONDARY OUTCOMES:
Adverse events of COVID-19 vaccines in cancer patients and health individuals | Up to 12 months
  Will use descriptive statistics (mean, median, range for continuous variables and frequency/percentage for categorical variables) to analyze demographic data including age, ethnicity, and comorbidity in healthy individuals and cancer patients as well as cancer type and current cancer treatment in cancer patients in association with adverse events after the vaccination.
T cell response to COVID-19 vaccine after vaccination in cancer patients and health individuals | Up to 12 months

OTHER OUTCOMES:
Incidence and severity of COVID-19 infection after the vaccination in cancer patients and health individuals | Up to 12 months
  Will use descriptive statistics (mean, median, range for continuous variables and frequency/percentage for categorical variables) to analyze demographic data including age, ethnicity, and comorbidity in healthy individuals and cancer patients as well as cancer type and current cancer treatment in cancer patients in association with incidence as well as severity of subsequent COVID-19 infection after the vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Saranya Chumsri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials